CLINICAL TRIAL: NCT02001766
Title: ATP Release and Sympathetic Nerve Activity in Patients With Type II Diabetes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anders Rasmussen Rinnov (Other)
Responsible Party: Sponsor-Investigator, Anders Rasmussen Rinnov, CIM administrator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-2-2011-070
Record Dates: First submitted 2013-11-19; First posted 2013-12-05 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes
Keywords: High intensity exercise; Glycemic control; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High intensity exercise (Experimental): 3 times per week in a total of 12 weeks
  Interventions: Behavioral: Exercise training
- Low intensity exercise (Experimental): 3 times per week in a total of 12 weeks
  Interventions: Behavioral: Exercise training
- Control (Experimental): Normal lifestyle for 12 weeks
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training

SUMMARY:
Type II diabetes (T2D) is characterized by endothelial dysfunction, resulting in a poor tissue perfusion and function as well as an increased risk of cardiovascular events. ATP, which is released from the red blood cells, contributes to the regulation of the blood flow and studies have shown that red blood cells taken from T2D patients have an impaired ability to release ATP. However, it is not known whether the changes in the ATP system is an underlying cause of the poor tissue perfusion observed in T2D. The purpose of project 1 is to test the hypothesis that the deterioration in blood flow in T2D is caused by a reduced release ATP from red blood cells, and to test if pharmacological manipulation of cAMP will normalize ATP release, plasma ATP levels and thereby blood flow.

Furthermore, epidemiological studies show a clear link between regular exercise and a reduced risk of serious cardiovascular disease. The extent to which a physically active lifestyle may improve endothelial function in T2D is unknown. Regular physical activity improves vascularization and induces an anti-inflammatory environment. Both the angiogenic and anti-inflammatory effects of physical activity is in part mediated by substances released from the active muscle. These muscle-derived substances are classified as myokines and have paracrine, autocrine and endocrine effects and may thereby affect distant tissues. The purpose of the project 2 is to investigate whether high intensity interval training may reverse endothelial dysfunction in T2D through increased release of ATP and myokines. In individuals with T2D we will determined blood flow in the muscle tissue using advanced ultrasound. In addition, using intravascular and intramuscular microdialysis we will determine ATP levels in blood and in the muscle interstitium.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetics
* BMI >30
* Non smokers
* Physical Inactive (less than 2 hours per week)

Exclusion Criteria:

* Thyroid disorder
* Known ischemic heart disease (intermittent claudication, angina)
* Diabetic eye disease
* Diabetic kidney disease
* Known heart disease
* Intake of beta-blockers
* Blood Pressure > 140/90
* Nephropathy and macroalbuminuria GFR measurement
* Acute illness within the last three weeks
* Chronic disease, including cancer, heart (ischemic and claudication), liver, kidney and respiratory disorders (asthma)
* Significant peripheral diabetic neuropathy (severe sensory disturbances)
* Significant peripheral diabetic angiopathy (former or current foot ulcer)
* Rheumatological disorders
* Pregnancy or childbirth within the past three months
* Alcohol abuse
* smokers
* Use of illegal performance-enhancing drugs (see IAAF list)
* Injuries and / or surgery within the last 6 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Glucose metabolism | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan P. Mortensen, Dr. Med., Study Chair — Centre of Inflammation and Metabolism
Locations (1):
- Centre of Inflammation and Metabolism (CIM), Rigshospitalet, Tagensvej 20, section M7641, Copenhagen, Denmark

REFERENCES:
- [Derived] Groen MB, Knudsen TA, Finsen SH, Pedersen BK, Hellsten Y, Mortensen SP. Reduced skeletal-muscle perfusion and impaired ATP release during hypoxia and exercise in individuals with type 2 diabetes. Diabetologia. 2019 Mar;62(3):485-493. doi: 10.1007/s00125-018-4790-0. Epub 2019 Jan 3. PMID 30607464